CLINICAL TRIAL: NCT03444519
Title: Brain Relaxation Facilitated by Mannitol in Craniotomy: Insight Into the Optimized Operation Window
Brief Title: The Therapeutic Time Window of Mannitol During Craniotomy for Optimal Brain Relaxation in Patients With Supratentorial Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, le tian wang, Principal Investigator, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KY2017-306
Record Dates: First submitted 2018-02-01; First posted 2018-02-23 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Supratentorial Tumors
Keywords: brain relaxation; mannitol; supratentorial tumours
MeSH Terms: conditions — Supratentorial Neoplasms | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol A (Experimental): in this group, Mannitol (1.0g/kg) is given just after the induction of general anesthesia
  Interventions: Drug: Mannitol
- Mannitol B (Active Comparator): in this group, Mannitol (1.0g/kg) is given at the time of skin incision
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Mannitol — This drug is in our routine use of neuroanesthesia, are given for facilitate brain relaxation

SUMMARY:
Although mannitol is used for brain relaxation during neurosurgery and in the treatment of raised intracranial pressure; there is not a consensus on its safe, effective dose and the duration of its administration. This study aimed to compare the effects of the mannitol in different use times, on the brain relaxation, electrolyte, lactate levels of the blood, peroperative fluid balance and the volume of the urine in supratentorial mass resection surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial shift >3mm
* Scheduled for supratentorial mass resection under elective conditions

Exclusion Criteria:

* Decompensated heart failure
* kidney insufficiency
* Diabetes insipidus,
* Electrolyte imbalance and
* Who are unconscious

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
brain relaxation score | just before dural opening
  difference in brain relaxation after drug administration
  The assessment was performed using a 4-point scale,
  1 denoting bulging or the condition that additional methods for brain relaxation are immediately and always required in order to continue the surgical procedure because of brain swelling;
  2, firm or the condition that additional methods for brain relaxation are occasionally required to continue the surgical procedure;
  3, adequate; 4, perfectly relaxed.
  In all patients, the degree of brain relaxation was assessed at the time of dural opening and satisfactory brain relaxation was defined as a brain relaxation score of 3 or 4.
  All the Secondary Outcome Measures below are observed the safety for intraoperative brain debulking during elective supratentorial craniotomy

SECONDARY OUTCOMES:
Blood sodium levels | change in 30 minute intervals in the first 2 hour after study drug administration
Blood potassium levels | change in 30 minute intervals in the first 2 hour after study drug administration
Blood chlorine levels | change in 30 minute intervals in the first 2 hour after study drug administration
Blood lactate levels | change in 30 minute intervals in the first 2 hour after study drug administration
Fluid balance during operation | change in 30 minute intervals in the first 2 hour after study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University affiliated Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided